CLINICAL TRIAL: NCT06174610
Title: Changes of Renal Resistive Index in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy - Observational Study.
Brief Title: Changes of Renal Resistive Index in Critically Ill Patients Undergoing Continuous Renal Replacement Therapy.
Status: Recruiting | Type: Observational
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Maciej Piwoda, Principal Investigator, Uniwersytecki Szpital Kliniczny w Opolu
Other Study IDs: RICRRT_USK
Record Dates: First submitted 2023-12-01; First posted 2023-12-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury (AKI); Continous Renal Replacement Therapy (CRRT); Critical Care; Renal Resistive Index (RRI)
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Kidney Injury + CRRT: Critically ill patients admitted to the intensive care unit (ICU), undergoing continuous renal replacement therapy due to Acute Kidney Injury.
  Diagnostic Test: Daily Doppler measurement of Renal Resistive Index
  Interventions: Diagnostic Test: Measurement of Renal Resistive Index

INTERVENTIONS:
Diagnostic Test: Measurement of Renal Resistive Index — The kidneys are preliminarily visualized in a 2D projection, followed by identifying interlobar or arcuate vessels using color Doppler. Flow measurements in these vessels are performed using pulsed-wave Doppler. Renal Resistive Index is determined over three cardiac cycles (five in the case of atrial fibrillation) in two different arteries, each in a different kidney section. Subsequently, measurements from each artery are averaged. If possible, the examination should be conducted bilaterally.
  The investigators do not have access to previous measurements (each study is recorded on a separate card).

SUMMARY:
The aim of the study is to determine whether there is a correlation between changes in the renal resistive index and the restoration of kidney function in critically ill patients undergoing continuous renal replacement therapy.

DETAILED DESCRIPTION:
A significant number of critically ill patients experience acute kidney injury (AKI), an independent factor contributing to increased mortality. Prevention of AKI and monitoring kidney function are crucial. Commonly used markers such as serum creatinine and hourly diuresis are employed to assess AKI severity, but they are not ideal due to their late elevation in the disease course. Therefore, alternative methods for detecting and evaluating kidney dysfunction at an earlier stage are sought.

Previous studies have demonstrated a correlation between the risk of AKI and the resistive index of renal parenchymal arteries. Renal resistive index (RRI) is a parameter calculated from Doppler measurements, representing the difference between peak blood velocity during systole and end-diastolic velocity divided by peak systolic velocity [(Vs-Vd) /Vs]. In healthy adult kidneys, the RI typically ranges from 0.6 to 0.7. Changes in RRI can be observed much earlier than an increase in serum creatinine concentration and/or a decrease in hourly diuresis.

Some patients with acute kidney injury require renal replacement therapy. Continuous renal replacement therapy (CRRT) is commonly used in critically ill patients, causing less circulatory destabilization compared to intermittent therapies. However, adverse effects accompany renal replacement therapies, including thromboembolic complications, bleeding, infections, blood cell damage, altered drug pharmacokinetics, and loss of proteins and vitamins.

In addition to determining the appropriate initiation time for CRRT, identifying the optimal moment to end the treatment is crucial. CRRT is typically applied for several days, and during the procedure, it is challenging to ascertain whether renal function has improved and whether CRRT can be safely discontinued. The hypothesis is that there may be a correlation between changes in RRI and the recovery of kidney function. This may enable the early identification of patients who have regained kidney function, allowing for the earlier termination of CRRT.

In 1989, a study was conducted on children undergoing peritoneal dialysis due to AKI, showing a relationship between a decrease in RRI and the restoration of kidney function. However, no similar study has been conducted on adult patients undergoing continuous renal replacement therapy.

The planned project will be based on daily ultrasonographic examinations, measuring RRI of the arcuate and/or interlobar arteries of both kidneys.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients undergoing CRRT due to AKI

Exclusion Criteria:

* age <18 years
* pregnancy
* history of chronic kidney disease in stage 4 or 5
* post-kidney transplant status
* mechanical circulatory support
* occurrence of one or more conditions preventing reliable RRI measurement in both kidneys:

  * challenging technical conditions of ultrasound examination, hindering proper visualization of the kidney
  * post-kidney injury in grade III and higher, according to AAST
  * advanced parenchymal kidney pathology: atrophy, hypoplasia, cirrhosis, extensive ischemia (more than 2/3 of the parenchyma),
  * kidney diseases preventing parenchyma identification: advanced cancer (stage above T1 according to TNM), certain forms of polycystic kidney disease
  * inflammatory kidney diseases
  * obstructive uropathy
  * renal vascular pathologies: renal vein thrombosis, significant stenosis (>60%), and renal artery occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients undergoing CRRT due to AKI
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-05-21 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Relationship between changes in RRI and recovery of kidney function | on average from 1 to 3 weeks
  The first ultrasound examination should be performed before the initiation of CRRT and, if not possible, within 24 hours of starting CRRT. Subsequently, the renal arteries will be assessed once a day during CRRT and after its completion until kidney function improves or there is a need for a return to renal replacement therapy. The return of kidney function is defined as a stable (increase <0.3 mg/dl/24h) or decreasing serum creatinine level in two consecutive tests conducted at intervals of at least 24 hours and an average hourly diuresis >0.5 ml/kg over the last 12 hours, with or without loop diuretics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Opole Voivodeship, Poland

REFERENCES:
- [Background] Patriquin HB, O'Regan S, Robitaille P, Paltiel H. Hemolytic-uremic syndrome: intrarenal arterial Doppler patterns as a useful guide to therapy. Radiology. 1989 Sep;172(3):625-8. doi: 10.1148/radiology.172.3.2672090.
- [Background] Katulka RJ, Al Saadon A, Sebastianski M, Featherstone R, Vandermeer B, Silver SA, Gibney RTN, Bagshaw SM, Rewa OG. Determining the optimal time for liberation from renal replacement therapy in critically ill patients: a systematic review and meta-analysis (DOnE RRT). Crit Care. 2020 Feb 13;24(1):50. doi: 10.1186/s13054-020-2751-8. PMID 32054522
- [Background] Fernandez SN, Santiago MJ, Gonzalez R, Lopez J, Solana MJ, Urbano J, Lopez-Herce J. Changes in hemodynamics, renal blood flow and urine output during continuous renal replacement therapies. Sci Rep. 2020 Nov 27;10(1):20797. doi: 10.1038/s41598-020-77435-x. PMID 33247145
- [Background] Fernandez SN, Lopez J, Gonzalez R, Solana MJ, Urbano J, Aguado A, Lancharro A, Lopez-Herce J, Santiago MJ. Doppler ultrasound in the assessment of renal perfusion before and during continuous kidney replacement therapy in the pediatric intensive care unit. Pediatr Nephrol. 2022 Dec;37(12):3205-3213. doi: 10.1007/s00467-022-05428-1. Epub 2022 Mar 14. PMID 35286455
- [Background] Ninet S, Schnell D, Dewitte A, Zeni F, Meziani F, Darmon M. Doppler-based renal resistive index for prediction of renal dysfunction reversibility: A systematic review and meta-analysis. J Crit Care. 2015 Jun;30(3):629-35. doi: 10.1016/j.jcrc.2015.02.008. Epub 2015 Feb 24. PMID 25746587